CLINICAL TRIAL: NCT06285409
Title: Comparing the Dose-response Profiles of Uterotonics After Initial Carbetocin Administration - an Ex-vivo Study in Desensitized Human Myometrium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-02
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Hemorrhage
Keywords: carbetocin; duratocin; oxytocin; uterine contraction
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin; Ergonovine; Carboprost; carboprost tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Carbetocin (Active Comparator): Dose-response testing with increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-5 M to 10-5 M
  Interventions: Drug: Carbetocin; Drug: Oxytocin
- Oxytocin (Active Comparator): Dose-response testing with increasing concentrations of oxytocin from 10-10 M to 10-5 M.
  Interventions: Drug: Carbetocin; Drug: Oxytocin
- Ergometrine (Active Comparator): Dose-response testing with increasing concentrations of ergometrine from 10-10 M to 10-5 M
  Interventions: Drug: Carbetocin; Drug: Oxytocin; Drug: Ergonovine
- Carboprost (Active Comparator): Dose-response testing with increasing concentrations of carboprost from 10-10 M to 10-5 M
  Interventions: Drug: Carbetocin; Drug: Oxytocin; Drug: Carboprost
- Control (Placebo Comparator): No drug added to physiological salt solution (PSS).
  Interventions: Drug: Carbetocin; Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin first bolus 10-8 M (equivalent to 100 mcg) will be added to the muscle bath to create ex-vivo environment similar to Cesarean delivery, and after 20 minutes the baths will be washed three time with physiological salt solution (PSS).
  Other Names: Duratocin
Drug: Oxytocin — Oxytocin 10-5M will be added to all strips for 2 hours to induce desensitization.
  Other Names: Pitocin
Drug: Carbetocin — Increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-5 M to 10-5 M
  Other Names: Duratocin
  Arms: Carbetocin
Drug: Oxytocin — Increasing concentrations of oxytocin from 10-10 M to 10-5 M
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Ergonovine — Increasing concentrations of ergometrine from 10-10 M to 10-5 M
  Other Names: Ergometrine
  Arms: Ergometrine
Drug: Carboprost — Increasing concentrations of carboprost from 10-10 M to 10-5 M
  Other Names: Hemabate
  Arms: Carboprost

SUMMARY:
This study will investigate the effects of drugs called "uterotonics" that help with the contraction of the uterus after a baby is born. This uterine contraction is very important to stop the bleeding after delivery. An uncontracted uterine state is called "uterine atony", which can lead to an excessive amount of post-delivery bleeding. Carbetocin is an uterotonic drug that works well to prevent post-delivery bleeding. In some cases, carbetocin is not enough to contract the uterus, and ongoing bleeding continues. When that happens, there are other uterotonic medications that can be used. In this study, we aim to find which uterotonic drug, amongst those available (oxytocin, carbetocin, ergometrine or carboprost), is more effective to lower the risk of post-delivery bleeding once carbetocin has already been administered.

This study will be done by using a very small sample of uterine tissue, taken from the incision site, following delivery by cesarean section. The sample is taken to the laboratory and will be exposed to carbetocin followed by other uterotonic drugs. The information obtained from this study will help modify the treatment for uterine atony and post-delivery bleeding to lower the risk further.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) remains to be one of the leading causes of maternal morbidity and mortality. It has been noted that an increasing number of PPH is attributed to the increased incidence of uterine atony. Carbetocin is the first line therapy for prevention and treatment of uterine atony. Carbetocin is currently used as a single dose treatment without an option of redosing. It has been proven that exposure to oxytocin during labour results in a decrease in myometrial contractions, previous studies shows that the current dose of carbetocin (100 µcg) is insufficient for optimal uterine contraction in failure to progress caesarean section.

According to current guidelines for medical management of PPH, the first line therapy for post CD uterotonic agent in Canada is carbetocin. It is a reliable and safe agent; however, it is a "one shot" option for treatment due to its longer half-life (40 minutes). The clinicians are reluctant to re-dose carbetocin after an initial failure to achieve adequate uterine tone with the assumption that the oxytocin receptors would likely be saturated with the agonist. It is unknown whether re-dosing with oxytocics (carbetocin or oxytocin) would help augment myometrial contractions, thereby lowering post-partum bleeding and improving patient outcomes. It is also unknown if prior carbetocin administration would affect myometrial contractility induced by other second line uterotonics such as ergometrine or carboprost.

This study is essential to answer the clinical question of the efficacy of re-dosing with either oxytocics or second line agents uterotonics following the first prophylactic dose of carbetocin in women with previously desensitized myometrium. This will help us better understand the comparative myometrial contractility response for a range of uterotonics.

The primary hypothesis of this study is that treating a second dose of oxytocics(carbetocin/oxytocin) in oxytocin pre-treated myometrium, after the first standard bolus of 100 µcg carbetocin will cause enhanced myometrial contraction compared to control.

The second hypothesis is that the efficacy of second line agents (ergometrine or carboprost) would not be as effective, i.e. they are likely to be less effective than oxytocics.

ELIGIBILITY:
Inclusion criteria

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring elective primary or first repeat CD
* Patients undergoing CD under spinal anesthesia

Exclusion criteria

* Patient refusal
* Patients who require general anesthesia
* Patients in labour and those receiving oxytocin for induction of labour
* Emergency CD
* placenta accreta spectrum disorder
* Patients who have had previous uterine surgery or >1 previous CD
* Patients with any condition predisposing to uterine atony and PPH (BMI > 40 kg/m2,
* Patients on medications that could affect myometrial contractility, such as insulin, nifedipine, labetalol or magnesium sulphate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Motility index | 4 hours
  Motility index (MI) is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  Frequency and amplitude are secondary outcome measures as described below.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 4 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 4 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist. The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No